CLINICAL TRIAL: NCT03272113
Title: Promoting Smoking Cessation During Pregnancy: a Combined Feasibility and Pilot Trial of a Theory-based Intervention Using Narrative, Images and Embedded Behaviour Change Techniques, Delivered Via Text-messaging
Brief Title: SKIP-IT Smoking Cessation in Pregnancy
Acronym: SKIP-IT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Stirling (Other)
Collaborators: Glasgow Caledonian University (Other); University of Dundee (Other); University of Southampton (Other); Edinburgh Napier University (Other)
Responsible Party: Principal Investigator, Helen Cheyne, Professor of Maternal and Child Health Research, University of Stirling
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: RMS2119; HIPS/16/4 (Other Grant/Funding Number: Scottish Government Chief Scientist Office)
Record Dates: First submitted 2017-08-29; First posted 2017-09-05 (Actual); Last update posted 2020-03-04 (Actual); Status verified 2020-03

CONDITIONS: Smoking Cessation; Pregnancy Related
MeSH Terms: conditions — Smoking Cessation

STUDY DESIGN:
Intervention Model Description: Behaviour change
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (No Intervention): Usual care to provided by smoking cessation services in the two study sites. Site one: support from a specialist advisor using motivational interviewing, one to one, group and telephone support.
  Site two: a smoking cessation incentive scheme administered through community pharmacies. Women who are verified by CO testing to have stopped smoking receive £12.50 per week.
- Intervention (Experimental): Women will receive usual care as described above plus the SKIP-IT intervention
  Interventions: Behavioral: SKIP-IT

INTERVENTIONS:
Behavioral: SKIP-IT — A theory-based intervention using narrative, images and embedded behaviour change techniques, delivered via text-messaging.
  Arms: Intervention

SUMMARY:
The aim of this study is to investigate the feasibility and likelihood of success of a narrative and image-based intervention, administered via text messages, for smoking cessation in pregnant women, prior to undertaking a large scale trial of its effectiveness. A feasibility and pilot trial will be undertaking involving 70 pregnant women who smoke in two NHS Boards.

DETAILED DESCRIPTION:
Smoking during pregnancy carries serious risks to mother and infant health. More babies whose mothers smoke are stillborn or die within the first year of life. Smoking during pregnancy results in increased rates of intrauterine growth retardation, preterm birth, and babies' longer-term risk of developing heart disease and diabetes. Pregnant women who smoke are more likely to experience miscarriage, placental abruption, pregnancy-induced hypertension and later conditions such as lung cancer and heart disease.

Reduction in smoking in pregnancy has been a long standing health policy target however there is limited evidence of effectiveness of many smoking cessation interventions and their uptake is generally low. We have developed, and carried out initial testing of an intervention to support smoking cessation in pregnant women using narrative, story-telling delivered via automated text-messages. The intervention aims to alter women's perceptions of risk, social norms, outcomes and self-efficacy using three key elements. 1. a narrative story of a fictional young pregnant woman 'Megan' trying to stop smoking by overcoming a series of commonplace barriers. 2) images showing the size of their fetus and its stage of development 3) an interactive 'help' function to receive a supportive, tailored response. Behaviour change techniques for smoking cessation in pregnancy are embedded in the intervention.

A randomised controlled trial is required to test the effectiveness of the intervention in reducing smoking in pregnancy. The aim of this study is to investigate the feasibility and likelihood of success of the narrative and image-based intervention for smoking cessation in pregnant women. If successful the intervention will be tested in a full-scale (Phase III) multi centre randomised controlled trial.

Objectives:

1. To assess acceptability and willingness to be randomised to the narrative and image based intervention or usual care.
2. To assess and compare the feasibility of recruitment strategies, the level of participants' retention in the study and engagement with the intervention.
3. To assess the acceptability and likely impact of the intervention among pregnant smokers.
4. To estimate the required sample size for a full trial.

ELIGIBILITY:
Inclusion Criteria:

1. Women 16 years of age or over,
2. Live within the catchment areas of study sites,
3. Up to and including 14 weeks of pregnancy,
4. Current smoker,
5. Own or regularly use a mobile phone with media capability,
6. Understand written English,
7. Able to give informed consent.

Exclusion Criteria:

1. Women who do not currently smoke,
2. Live outside the catchment areas of study sites,
3. Over 14 weeks of pregnancy,
4. Do not use or have access to a mobile phone with media capability,
5. Cannot understand written English,
6. Not able to give informed consent,
7. Already enrolled in an alternative formal smoking cessation trial at the time of referral to the study.

Min Age: 16 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2017-12-05 (Actual); Primary Completion 2018-10-16 (Actual); Study Completion 2019-08-31 (Actual)

PRIMARY OUTCOMES:
Recruitment rate | 23 months
  Progression to a full trial will require recruitment ≥50% of women who give permission to have their details passed to the research team (i.e. those who express initial interest in the study).
Drop out rate | 23 months
  Progression to a full trial will require <30% dropout
Direction of effect | 23 months
  Progression to a full trial will require direction of effect on smoking cessation rate in favour of the intervention.

SECONDARY OUTCOMES:
Engagement | 23 months
  Engagement in the intervention will be assessed using data captured by the computer system which monitors the text message responses.
Acceptability | 23 months
  Acceptability of the intervention will be assessed in short interviews conducted with intervention group participants at the follow-up points

OTHER OUTCOMES:
Smoking cessation outcomes | At each subsequent data collection time-point (4 weeks post-randomisation, 36 weeks of pregnancy, 6-7 weeks post due-date, 12-13 weeks post due-date)
  1. The Russell Standard abstinence question: if they have smoked at all since the last data collection point (with answers being reported as: 'no, not a puff; 1-5 cigarettes; more than 5 cigarettes'). [self-reported abstinence]
  2. How many times they have purposefully not smoked for more than 24 hrs since the last data collection time point. [Self-reported 24hr quit attempts]

CONTACTS AND LOCATIONS:
Locations (2):
- United Kingdom (2):
  - NHS Ayrshire and Arran, Ayr
  - NHS Tayside, Perth